CLINICAL TRIAL: NCT01815164
Title: Effect of Hypnotherapy and Educational Intervention on Brain Response to Visceral Stimulus Perception in the Irritable Bowel Syndrome
Brief Title: Effect of Hypnotherapy and Educational Intervention in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Mats Lowén, MD, University Hospital, Linkoeping
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M71-09
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnotherapy (Active Comparator): Hypnotherapy
  Interventions: Behavioral: Hypnotherapy
- Educational intervention (Active Comparator): Educational intervention
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Hypnotherapy — Gut-directed hypnotherapy administered by an experienced hypnotherapist.
  Arms: Hypnotherapy
Behavioral: Educational intervention — Educational intervention vith education regarding Irritabel bowel Syndrome.
  Arms: Educational intervention

SUMMARY:
Aim: Gut directed hypnotherapy can reduce IBS symptoms but the mechanisms underlying this therapeutic effect remain unknown. We determined the effect of hypnotherapy and educational intervention on brain responses to cued rectal distensions in IBS patients. Methods: 44 women with moderate to severe IBS and 20 healthy controls (HCs) were included.. Blood oxygen level dependent (BOLD) signals were measured by functional Magnetic Resonance Imaging (fMRI) during expectation and delivery of high (45 mmHg) and low (15 mmHg) intensity rectal distensions. Twenty-five patients were assigned to hypnotherapy (HYP) and 16 to educational intervention (EDU). 31 patients completed the treatments and the post treatment fMRI. Results: Similar symptom reduction was achieved in both groups. HYP responders demonstrated a pre-post treatment BOLD attenuation in both anterior and posterior insula during high intensity distension, while EDU responders had a BOLD attenuation in prefrontal cortex. Pre-post differences for the low distension and for the two expectation conditions were almost exclusively seen in the HYP group. For all responders there was a significant correlation between treatment induced reduction of GI related anxiety and BOLD decrease in the anterior insula. Following treatment, the brain response to distension was similar to that observed in HCs, suggesting that the treatment had a normalizing effect on the central processing abnormality of visceral signals in IBS. Conclusions: The abnormal processing and enhanced perception of visceral stimuli in IBS can be normalized by psychological interventions. Symptom improvement in the treatment groups may be mediated by different brain mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Rome III Female Age 20-60 Swedish speaking Right-handed

Exclusion Criteria:

Central acting medication IBD Psychiatric diseases Abdominal surgery NictoinePacemaker Prosthesis Metal in the brain Claustrophobia Large tattoo

-

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Walter, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- University Hospital, Linköping, Sweden

REFERENCES:
- [Background] Larsson MB, Tillisch K, Craig AD, Engstrom M, Labus J, Naliboff B, Lundberg P, Strom M, Mayer EA, Walter SA. Brain responses to visceral stimuli reflect visceral sensitivity thresholds in patients with irritable bowel syndrome. Gastroenterology. 2012 Mar;142(3):463-472.e3. doi: 10.1053/j.gastro.2011.11.022. Epub 2011 Nov 19. PMID 22108191
- [Derived] Lowen MB, Mayer EA, Sjoberg M, Tillisch K, Naliboff B, Labus J, Lundberg P, Strom M, Engstrom M, Walter SA. Effect of hypnotherapy and educational intervention on brain response to visceral stimulus in the irritable bowel syndrome. Aliment Pharmacol Ther. 2013 Jun;37(12):1184-97. doi: 10.1111/apt.12319. Epub 2013 Apr 25. PMID 23617618